CLINICAL TRIAL: NCT00445692
Title: Maintenance Therapy With Lenalidomide, Dexamethasone and Clarithromycin (Biaxin) Following Autologous/Syngeneic Transplant for Multiple Myeloma
Brief Title: Lenalidomide, Dexamethasone, and Clarithromycin in Treating Patients Who Have Undergone Stem Cell Transplant for Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Leona Holmberg, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2135.00; NCI-2010-02116 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2135.00p; 2135; 2135.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Results first posted 2018-03-21 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: DS Stage I Plasma Cell Myeloma; DS Stage II Plasma Cell Myeloma; DS Stage III Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Clarithromycin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (clarithromycin, dexamethasone, lenalidomide) (Experimental): Patients receive clarithromycin orally (PO) twice daily and dexamethasone PO once a week. Treatment with clarithromycin and dexamethasone continues for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also receive lenalidomide PO once daily on days 1-14. Courses with lenalidomide repeat every 21 days in the absence of disease progression or unacceptable toxicity. Lenalidomide is taken 4 hours or more after last dose of daily clarithromycin.
  NOTE: *After one year of treatment, dexamethasone is tapered for an additional 4 weeks.
  Interventions: Drug: Clarithromycin; Drug: Dexamethasone; Drug: Lenalidomide

INTERVENTIONS:
Drug: Clarithromycin — Given Orally (PO)
  Other Names: Abbott-56268; Biaxin
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Lenalidomide — Given Orally (PO)
  Other Names: CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This phase II trial studies lenalidomide, dexamethasone, and clarithromycin in treating patients who have undergone stem cell transplant for multiple myeloma. Biological therapies, such as lenalidomide and clarithromycin, may stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving lenalidomide together with dexamethasone and clarithromycin may be an effective treatment for multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the toxicity of the use of lenalidomide/biaxin (clarithromycin)/dexamethasone as maintenance therapy after autologous/syngeneic transplant.

II. Evaluate the median time to disease progression. III. Evaluate survival.

OUTLINE:

Patients receive clarithromycin orally (PO) twice daily (BID) and dexamethasone PO once a week. Treatment with clarithromycin and dexamethasone continues for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also receive lenalidomide PO once daily (QD) on days 1-14. Courses with lenalidomide repeat every 21 days in the absence of disease progression or unacceptable toxicity.

NOTE: *After one year of treatment, dexamethasone is tapered for an additional 4 weeks.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Any autologous or syngeneic patient who underwent high dose melphalan (>= 140 mg/m^2) therapy/peripheral blood stem cell (PBSC) or bone marrow (BM) rescue for any stage of multiple myeloma and did not participate in another clinical transplant trial which is also evaluating long-term disease free survival or survival
* Platelet count (transfusion independent) > 50,000 cells/mm^3 and absolute granulocyte count > 1500 cells/mm^3 for 5 calendar days after recovery from high dose therapy
* Patients should be between 30 days to 120 days after transplant
* Willingness and ability to comply with Food and Drug Administration (FDA)-mandated REV ASSIST Program, Celgene System for Lenalidomide Education and Prescribing Safety
* Signing a written informed consent form

Exclusion Criteria:

* Karnofsky score less than 70
* A left ventricular ejection fraction less than 45% immediately pre transplant; patients with congestive heart disease with transplant, history of myocardial infarction (MI), or history of coronary artery disease
* Total bilirubin greater than 2 mg/ml (unless history of Gilbert's disease), serum glutamic-oxaloacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) > 2.5 x upper limit of normal
* Calculated by Cockcroft-Gault formula or measured serum creatinine clearance < 25 ml/minute
* Pregnant and/or lactating females
* Patients who cannot give informed consent
* Patients with untreated systemic infection
* Patients with history prior to transplant of treatment with combination therapy Lenalidomide/Biaxin and steroid without response
* Patients allergic to lenalidomide, biaxin or dexamethasone
* Referring physician not registered with REV ASSIST program or unwilling to oversee the care of the patients on study and comply with the FDA-mandated REV ASSIST Program
* Patients unwilling to practice adequate forms of contraception if clinically indicated until 30 days after stopping therapy; male patients on study need to be consulted to use latex condoms (even if they have had a vasectomy) every time they have sex with a woman who is able to have children while they are being treated and for 30 days after stopping drugs
* Patients with >= grade 3 peripheral neuropathy
* Prior history of uncontrollable side effects to dexamethasone therapy
* A prior history of human immunodeficiency virus (HIV) positivity with pre-transplant evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-01-10 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona Holmberg, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 32 patients were enrolled. 31 patients started therapy. 1 patient was consented but was deemed ineligible prior to therapy initiation.
Groups:
- Treatment (Clarithromycin, Dexamethasone, Lenalidomide): Patients receive clarithromycin orally twice daily and dexamethasone orally once a week. Treatment with clarithromycin and dexamethasone continues for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also receive lenalidomide orally once daily on days 1-14. Courses with lenalidomide repeat every 21 days in the absence of disease progression or unacceptable toxicity. Lenalidomide is taken 4 hours or more after last dose of daily clarithromycin.
  NOTE: *After one year of treatment, dexamethasone is tapered for an additional 4 weeks.
  Clarithromycin: Given Orally (PO)
  Dexamethasone: Given PO
  Lenalidomide: Given PO
Period: Overall Study
Arm/Group | Treatment (Clarithromycin, Dexamethasone, Lenalidomide)
Started | 31
Completed | 15
Not Completed | 16
Not completed — Adverse Event | 11
Not completed — Lack of Efficacy | 5

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Clarithromycin, Dexamethasone, Lenalidomide): Patients receive clarithromycin orally (PO) twice daily and dexamethasone PO once a week. Treatment with clarithromycin and dexamethasone continues for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also receive lenalidomide PO once daily on days 1-14. Courses with lenalidomide repeat every 21 days in the absence of disease progression or unacceptable toxicity. Lenalidomide is taken 4 hours or more after last dose of daily clarithromycin.
  NOTE: *After one year of treatment, dexamethasone is tapered for an additional 4 weeks.
  Clarithromycin: Given Orally (PO)
  Dexamethasone: Given PO
  Lenalidomide: Given PO
Arm/Group | Treatment (Clarithromycin, Dexamethasone, Lenalidomide)
Number analyzed (Participants) | 31
Age, Continuous [Mean (Full Range); unit: years] — Age at transplant
  years | 58 [28 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 28
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Episodes of Grade 3-4 Non Infectious, Non-dermatological or Non-neurological Toxicities, Episodes of Any Infections, Grade 3-4 Dermatological or Episodes of Grade 2-3 Peripheral Neuropathy Common Terminology Criteria for Adverse Events Version 3
Time Frame: First year of therapy
Measure: Number; unit: episodes
Groups:
- Treatment (Clarithromycin, Dexamethasone, Lenalidomide): Patients receive clarithromycin orally (PO) twice a day and dexamethasone PO once a week. Treatment with clarithromycin and dexamethasone continues for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also receive lenalidomide PO daily on days 1-14. Courses with lenalidomide repeat every 21 days in the absence of disease progression or unacceptable toxicity. Lenalidomide is taken 4 hours or more after last dose of daily clarithromycin.
  NOTE: *After one year of treatment, dexamethasone is tapered for an additional 4 weeks.
  Clarithromycin: Given PO
  Dexamethasone: Given PO
  Lenalidomide: Given PO
Arm/Group | Treatment (Clarithromycin, Dexamethasone, Lenalidomide)
Number analyzed (Participants) | 31
episodes
  Neutropenia | 6
  Thrombocytopenia | 1
  Deep venous thrombus/Pulmonary Embolism | 1
  Anemia | 1
  Pneumonia | 4
  Upper respiratory infections | 12
  Sinusitis/acute otitis media | 3
  Epiglottic appendagitis | 1
  Cellulitis | 3
  Clostridium difficile colitis | 1
  Vaginitis | 3
  Peripheral neuropathy | 10
  Dermal leukocytic vasculitis | 1
  Secondary cancer Acute Myeloid Leukemia | 1
  Re-occurrence of skin cancer | 1

2. Primary Outcome: Time to Disease Progression
Description: International Myeloma Working Group Uniform Response Criteria was used
Time Frame: Up to 10.25 years
Population: Measured among the 20 patients who progressed
Measure: Median (Full Range); unit: months
Groups:
- Treatment (Clarithromycin, Dexamethasone, Lenalidomide): Patients receive clarithromycin PO BID and dexamethasone PO once a week. Treatment with clarithromycin and dexamethasone continues for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also receive lenalidomide PO QD on days 1-14. Courses with lenalidomide repeat every 21 days in the absence of disease progression or unacceptable toxicity. Lenalidomide is taken 4 hours or more after last dose of daily clarithromycin.
  NOTE: *After one year of treatment, dexamethasone is tapered for an additional 4 weeks.
  Clarithromycin: Given PO
  Dexamethasone: Given PO
  Lenalidomide: Given PO
Arm/Group | Treatment (Clarithromycin, Dexamethasone, Lenalidomide)
Number analyzed (Participants) | 20
months | 30.5 [15 to 68.4]

3. Secondary Outcome: Survival
Description: number of patients alive or dead
Time Frame: From date of transplant until the date of death from any cause, assessed up to 10.25 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Clarithromycin, Dexamethasone, Lenalidomide)
Number analyzed (Participants) | 31
Participants
  Multiple meyloma deaths | 10
  Acute Myeloid Leukemia death | 1
  Lung cancer death | 1
  Heart attack death | 1
  Alive | 18

ADVERSE EVENTS:
Time Frame: 10.25 years
Arm/Group | Treatment (Clarithromycin, Dexamethasone, Lenalidomide)
All-Cause Mortality (participants affected / at risk) | 13/31
Serious Adverse Events (participants affected / at risk) | 11/31
Other Adverse Events (participants affected / at risk) | 19/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Clarithromycin, Dexamethasone, Lenalidomide) (N=31)
Upper Respiratory Syncytial Virus infection (Infections and infestations) | 1
Varicella-zoster virus pneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Peripheral edema (Cardiac disorders) | 1
Pneumocystis Carinii Pneumonia (Infections and infestations) | 1
H1N1 influenza / Streptococcus pneumonia (Infections and infestations) | 1
Ileus (Gastrointestinal disorders) | 1
Secondary cancer, Acute Myeloid Leukemia (Blood and lymphatic system disorders) | 1
Upper respiratory syncytial viurs infection/Leukocytoclastic vasculitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Clarithromycin, Dexamethasone, Lenalidomide) (N=31)
Peripheral Neuropathy (Nervous system disorders) | 10 — grades 2 and 3 only occurred
Neutropenia (Investigations) | 9 — grades 2-4 reported, grade 2 ( n=3) , grade 3 (n=4), grade 4 (n=2).
upper respiratory infection (Infections and infestations) | 11
sinus/acute otitis (Infections and infestations) | 3
cellulitis (Infections and infestations) | 3
vaginitis (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-10-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT00445692/Prot_SAP_000.pdf